CLINICAL TRIAL: NCT02269722
Title: A Comparison of Radial Artery Clamp Times in Patients Undergoing Cardiac Catheterization Via a Percutaneous Transradial Approach
Brief Title: Postcath Radial Arterial Clamp Time In the CAth Lab
Acronym: PRACTICAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shahar Lavi, Interventional Cardiologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10796
Record Dates: First submitted 2014-09-28; First posted 2014-10-21 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short Clamp time (Experimental): Radial clamp applied at full pressure for 20 minutes. At the end of 20 minutes, the clamp will be loosened ¼ turn every 5 minutes over 20 minutes and then removed.
  Interventions: Device: Vascular compression device- RADAR TM-Short clamp time
- Long Clamp Time (Experimental): Radial clamp applied at full pressure for 60 minutes. At the end of 60 minutes, the clamp is to be loosened and removed under the same instruction as those patients in arm one.
  Interventions: Device: Vascular compression device RADAR TM-Long clamp time

INTERVENTIONS:
Device: Vascular compression device- RADAR TM-Short clamp time — A clamp is placed on the radial artery following cardiac catheterization for 20 minutes
  Arms: Short Clamp time
Device: Vascular compression device RADAR TM-Long clamp time — A clamp is placed on the radial artery following cardiac catheterization for 20 minutes
  Arms: Long Clamp Time

SUMMARY:
The investigators will assess the effect of different times of radial clamp post procedure on radial artery occlusion and bleeding.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety of shorter radial artery clamp time post cardiac catheterization with respect to achieving hemostasis and the incidence of radial artery occlusion. The investigators hypothesize that shorter radial artery clamp times following cardiac catheterization will achieve similar hemostasis to longer clamp times with a decrease in the incidence of radial artery occlusion.

ELIGIBILITY:
Inclusion Criteria:

* All patients who require cardiac catheterization via the radial approach for the investigation and treatment of coronary artery disease.
* Patients must have evidence of pre-procedural radial artery patency using Barbeau test.
* Patients must be able to give informed consent

Exclusion Criteria:

* Evidence of pre-procedural radial artery thrombosis
* Inability to give informed consent
* Patient desire not to participate in the study
* Emergent procedures when the delay associated for obtaining informed consent may affect patient outcome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Incidence of radial artery occlusion | 24 hours
  Flow assessed by pulse oximeter

SECONDARY OUTCOMES:
Bleeding | 24 hours
  Need to retighten clamp, ooze, hematoma

CONTACTS AND LOCATIONS:
Overall Officials: Shahar Lavi, MD, Principal Investigator — LHSC
Locations (1):
- London Health Science Center, London, Ontario, Canada

REFERENCES:
- [Derived] Lavi S, Cheema A, Yadegari A, Israeli Z, Levi Y, Wall S, Alemayehu M, Parviz Y, Murariu BD, McPherson T, Syed J, Bagur R. Randomized Trial of Compression Duration After Transradial Cardiac Catheterization and Intervention. J Am Heart Assoc. 2017 Feb 3;6(2):e005029. doi: 10.1161/JAHA.116.005029. PMID 28159821